CLINICAL TRIAL: NCT02942199
Title: MySafeRx & MedicaSafe Open-Label Buprenorphine Induction and Lapse Evaluation (MyMOBILE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Collaborators: MedicaSafe, Inc. (Industry); MySafeRx, Inc (Unknown); Dartmouth College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHA-IRB-1029/03/16
Record Dates: First submitted 2016-10-20; First posted 2016-10-24 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MySafeRx Intervention (Experimental): The MySafeRx platform is a combination of several key components, including daily videoconferencing check-ins with motivational interviewing-based recovery coaching, text-messaging reminders, secure storage of buprenorphine medication within a secure electronic pill dispenser, and a standardized protocol for supervising self-administration of medication via videoconferencing. This arm represents MySafeRx using the MedicaSafe 3000 electronic pill dispenser.
  Interventions: Other: MySafeRx

INTERVENTIONS:
Other: MySafeRx — The MySafeRx platform is a combination of several key components, including daily videoconferencing check-ins with motivational interviewing-based recovery coaching, text-messaging reminders, secure storage of buprenorphine medication within a secure electronic pill dispenser (i.e., MedicaSafe 3000), and a standardized protocol for supervising self-administration of medication via videoconferencing.

SUMMARY:
The goal of the MyMOBILE study is to evaluate the feasibility, acceptability, and usability of a novel platform that integrates text messaging reminders, secure electronic pill organizers, and daily remote brief motivational recovery support visits with a standardized protocol for supervised self-administration of buprenorphine via videoconferencing.

DETAILED DESCRIPTION:
Opioid use disorder is a serious public health issue. Buprenorphine/ Naloxone (B/N) is a partial opioid mu-receptor agonist dosed daily that prevents opioid withdrawal, blocks opioid euphoria and can prevent opioid overdose. Extended treatment with B/N increases rates of abstinence and outpatient treatment retention and decreases Hepatitis C (HCV) transmission. B/N treatment dropout is associated with relapse and overdose death.

B/N adherence may be a critical factor influencing retention and reducing overall healthcare costs. Also, B/N diversion is associated with poor adherence and has become increasingly common and worrisome. While many patients achieve stability after starting B/N treatment, more than 80% of 18-25 year olds leave treatment within a year with relapse as the most common reason. Ongoing illicit opioid use during treatment increases odds of relapse and dropout. The MySafeRx platform helps prescribers offer a higher level of support for vulnerable patients with opioid use disorder during periods of clinical instability. The MySafeRx platform is a combination of several key components, including daily videoconferencing check-ins with motivational interviewing-based recovery coaching, text-messaging reminders, secure storage of B/N medication within a secure electronic pill dispenser, and a standardized protocol for supervising self-administration of medication via videoconferencing. By offering this recovery support and medication adherence monitoring program during periods of instability, this system could improve treatment outcomes by ensuring increased adherence, while also preventing B/N diversion.

This study primarily seeks to demonstrate the feasibility of the MySafeRx platform among young adults (18-39 years, inclusive) with opioid use disorders. While each key component may have an individual therapeutic effect, the investigators hypothesize that an integrated process involving all key components may be necessary to unlock the full therapeutic potential of a mobile platform for daily remote supervised self-administration and diversion prevention among this group. Providing targeted motivational interviewing and recovery support at this context-specific moment of daily medication-taking when people are very receptive to treatment may offer a new opportunity for expanding how recovery support can be delivered.

This study will enroll patients (18-39 years old) in office-based opioid treatment currently prescribed buprenorphine by a CHA prescriber who had illicit-opioid positive urine screens in the past week or who have just received buprenorphine induction. We will start participants with MySafeRx using the MedicaSafe 3000 dispenser and will assess for feasibility, acceptability, and usability during a 30 day period. Assessments will be conducted at baseline, two and four weeks.

ELIGIBILITY:
Inclusion Criteria:

Participants must:

1. Be between the ages of 18 and 39 years old.
2. Be able to provide informed consent.
3. Be clinically diagnosed with opioid dependence (DSM-IV) or opioid use disorder (DSM-5).
4. Be currently in Medication-Assisted Treatment (MAT) with buprenorphine.
5. Test positive for illicit opioid use within the past week.
6. Have an Android smartphone or tablet device with current access to the internet through secure WiFi and/or a mobile data plan.
7. Be able to meet in a confidential place for scheduled videoconferencing call with Mobile Recovery Coach on a daily basis.

Exclusion Criteria:

Participants must not:

1. Be younger than 18 or older than 39 years of age.
2. Be non-English speaking.
3. Be otherwise unable to complete informed consent.
4. Be in their third trimester of pregnancy.
5. Have cognitive deficits that may limit their ability to complete study procedures.
6. Receive a twice daily prescription of buprenorphine.
7. Exhibit use of an illicit substance or prescribed medication considered by the PI to be unsafe for use with the MySafeRx device or study procedures.
8. Exhibit signs of severe mental illness such as psychoses, present with active suicidal ideation, or otherwise be a risk to themselves or others.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Adherence | 4 weeks
  Feasibility will be measured by percentage of study days with confirmation of supervised self-administration of medication.
Usability | 2 weeks, 4 weeks
  Level of patient usability as measured by system usability scale
Acceptability | 4 weeks
  Level of patient acceptability of system

CONTACTS AND LOCATIONS:
Overall Officials: Zev Schuman-Olivier, Principal Investigator — Cambridge Health Alliance; Harvard Medical School
Locations (1):
- Cambridge Health Alliance, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schuman-Olivier Z, Weiss RD, Hoeppner BB, Borodovsky J, Albanese MJ. Emerging adult age status predicts poor buprenorphine treatment retention. J Subst Abuse Treat. 2014 Sep;47(3):202-12. doi: 10.1016/j.jsat.2014.04.006. Epub 2014 May 20. PMID 24953168
- [Background] Schuman-Olivier Z, Borodovsky JT, Steinkamp J, Munir Q, Butler K, Greene MA, Goldblatt J, Xie HY, Marsch LA. MySafeRx: a mobile technology platform integrating motivational coaching, adherence monitoring, and electronic pill dispensing for enhancing buprenorphine/naloxone adherence during opioid use disorder treatment: a pilot study. Addict Sci Clin Pract. 2018 Sep 24;13(1):21. doi: 10.1186/s13722-018-0122-4. PMID 30249279
- See also: Website for Cambridge Health Alliance Institutional Review Board — http://www.challiance.org/academic/institutional-review-board.aspx
- See also: Website for Cambridge Health Alliance Outpatient Addictions Service — http://www.challiance.org/cha-services/outpatient-addictions-service.aspx
- See also: Website for MedicaSafe 3000 — http://www.medicasafe.com